CLINICAL TRIAL: NCT04407832
Title: A Double Blind Study Comparing Low Dose and High Dose IV Esomeprazole After Successful Endoscopic Therapy in Patients With Peptic Ulcer Bleeding
Brief Title: Comparing Two Doses of IV Esomeprazole After Successful Endoscopic Therapy
Acronym: lowdosePPI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Collaborators: Taipei Medical University Hospital (Other); Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: lowdosePPI
Record Dates: First submitted 2011-08-04; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Peptic Ulcer Bleeding
Keywords: hemostasis; heat probe; hemoclip; rebleeding
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose PPI (Active Comparator): 40 mg esomeprazole IV for three days followed by esomeprazole 40 mg po daily for two months
  Interventions: Device: heat probe or hemoclip
- high dose PPI (Active Comparator): 40 mg esomeprazole IV every 6 hr for 3 days followed by 40 mg po daily for two months
  Interventions: Device: heat probe or hemoclip

INTERVENTIONS:
Device: heat probe or hemoclip — for hemostasis
  Other Names: Olympus co.
  Arms: low dose PPI
Device: heat probe or hemoclip — for hemostasis
  Other Names: Olympus co.
  Arms: high dose PPI

SUMMARY:
The investigators used two different doses of esomeprazole (40 mg IV q.d. and 40 mg IV q6h for three days followed by esomeprazole 40 mg q.d. orally in two groups) after successful endoscopic therapy with heat probe therapy or hemoclip placement.

The goal of this study is to assess the outcomes of two different regimens of low vs. high dose of intravenous esomeprazole after endoscopic therapy in patients with peptic ulcer bleeding.

DETAILED DESCRIPTION:
A bleeding peptic ulcer remains a serious medical problem with significant morbidity and mortality. Endoscopic therapy significantly reduces further bleeding, surgery, and mortality in patients receiving intravenous Proton Pump Inhibitor (PPI）and is now recommended as the first hemostatic modality for these patients. In the past few years, adjuvant use of a high-dose proton pump inhibitor (PPI) after endoscopic therapy has been endorsed in some studies, including two consensus statements and two meta-analysis. To sustain a high intragastric pH, a high dose of omeprazole has been used in previous studies concerning high-risk peptic ulcer bleeding. However, in one recent published metaanalysis found that low dose PPI may be as effective as high dose PPI in preventing further bleeding in high-risk patients. Therefore, one double blind study is needed clarify this puzzle.

We used two different doses of esomeprazole (40 mg IV q.d. and 40 mg IV q6h for three days followed by esomeprazole 40 mg q.d. orally in two groups) after successful endoscopic therapy with heat probe therapy or hemoclip placement.

The goal of this study is to assess the outcomes of two different regimens of low vs. high dose of intravenous esomeprazole after endoscopic therapy in patients with peptic ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

* patients with peptic ulcer bleeding with active bleeding or nonbleeding visible (initial Hb<10, shock, or coffee grounds or blood in stomach)

Exclusion Criteria:

* age >90y/o
* pregnant woman
* allergic to esomeprazole
* unwilling to enter this study
* bleeding tendency
* severe co-morbid illness, including cancer, hepatic failure, renal failure,

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
further bleeding | 14 days
  Number of participants with rebleeding within 14 days

SECONDARY OUTCOMES:
hospital stay | 30 days
  hospital stay in day
need of blood transfusion | 30 days
  number of participants need of blood transufion
surgical intervention | 30 days
  number of participants need surgical intervention to manage bleeding
mortality | 30 days
  number of participants death

CONTACTS AND LOCATIONS:
Overall Officials: Hwai-jeng Lin, M.D., Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Division of Gastroenterology, TMUH, Taipei, Taiwan